CLINICAL TRIAL: NCT00283959
Title: A Phase 2, Open-Label, Single Dose Level, 12-Week Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of AT1001 in Patients With Fabry Disease
Brief Title: A 12-Week Safety and Pharmacodynamic Study of AT1001 (Migalastat Hydrochloride) in Participants With Fabry Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAB-CL-202 (AA1565521)
Record Dates: First submitted 2006-01-27; First posted 2006-01-31 (Estimated); Results first posted 2018-09-07 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Fabry Disease
Keywords: Amicus Therapeutics; AT1001; Galafold; Migalastat; Substrate
MeSH Terms: conditions — Fabry Disease | interventions — migalastat; larazotide acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Migalastat (Experimental): Migalastat 150 mg was administered orally QOD during the 12-week treatment period and then during the optional 36-week extension period.
  Interventions: Drug: migalastat HCl

INTERVENTIONS:
Drug: migalastat HCl
  Other Names: AT1001; Galafold; migalastat

SUMMARY:
Study to evaluate the safety, tolerability, and pharmacodynamics of migalastat hydrochloride (HCl) (migalastat) and how migalastat works in participants with Fabry disease.

DETAILED DESCRIPTION:
This was a Phase 2, open-label study in male participants with Fabry disease. The study consisted of a 4-week screening period during which participants' genotype was assessed for α-galactosidase A (α-Gal A) activity in response to migalastat via an in vitro assay. Participants were required to have α-Gal A activity responsive to migalastat. The study consisted of a 12-week treatment period, followed by an optional 36-week extension period. Participants received migalastat 150 milligrams (mg) once every other day (QOD) for 12 weeks during the treatment period. Participants could then opt to participate in the extension period.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18 and 65 years of age (inclusive)
* Hemizygous for Fabry disease
* Had a confirmed diagnosis of Fabry disease with a documented missense gene mutation (individual or familial)
* Had enhanceable enzyme activity based on in vitro tests
* Had documented evidence of cardiac and/or renal dysfunction (for example, abnormal electrocardiogram (ECG), left ventricular hypertrophy, renal insufficiency) and/or cerebral tissue dysfunction documented by evidence of stroke and/or peripheral nervous tissue dysfunction (for example, intolerance to heat/cold, decrease of perspiration)
* Must have been previously untreated by enzyme replacement therapy (ERT) or substrate depletion for Fabry disease or were able to stop ERT for at least 18 weeks or up to three months, and be willing to undergo two kidney and three skin biopsies
* Agreed to be sexually abstinent or use a condom with spermicide when engaging in sexual activity during the course of the study and for a period of 30 days following their completion of the study
* Were willing and able to sign an informed consent form

Exclusion Criteria:

* History of significant disease other than Fabry disease
* History of organ transplant
* Serum creatinine >2 mg per deciliter on Day -2
* Screening 12-lead ECG demonstrating corrected QT interval >450 milliseconds prior to dosing
* Pacemaker or other contraindication for magnetic resonance imaging (MRI) scanning
* Took any of the following prohibited medications: Fabrazyme® (agalsidase beta), Replagal™ (agalsidase alfa), Glyset® (miglitol), Zavesca® (miglustat), or any experimental therapy for any indication
* Participated in a previous clinical trial in the last 30 days
* Any other condition, which, in the opinion of the investigator, would jeopardize the safety of the participant or impact the validity of the study results

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-06-27 (Actual); Primary Completion 2008-05-08 (Actual); Study Completion 2008-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Clinical Research, Study Director — Amicus Therapeutics
Locations (2):
- Parkville, Australia
- Porto Alegre, Brazil

REFERENCES:
- [Derived] Benjamin ER, Della Valle MC, Wu X, Katz E, Pruthi F, Bond S, Bronfin B, Williams H, Yu J, Bichet DG, Germain DP, Giugliani R, Hughes D, Schiffmann R, Wilcox WR, Desnick RJ, Kirk J, Barth J, Barlow C, Valenzano KJ, Castelli J, Lockhart DJ. The validation of pharmacogenetics for the identification of Fabry patients to be treated with migalastat. Genet Med. 2017 Apr;19(4):430-438. doi: 10.1038/gim.2016.122. Epub 2016 Sep 22. PMID 27657681
- [Derived] Germain DP, Giugliani R, Hughes DA, Mehta A, Nicholls K, Barisoni L, Jennette CJ, Bragat A, Castelli J, Sitaraman S, Lockhart DJ, Boudes PF. Safety and pharmacodynamic effects of a pharmacological chaperone on alpha-galactosidase A activity and globotriaosylceramide clearance in Fabry disease: report from two phase 2 clinical studies. Orphanet J Rare Dis. 2012 Nov 24;7:91. doi: 10.1186/1750-1172-7-91. PMID 23176611

RESULTS

PARTICIPANT FLOW:
Groups:
- Migalastat: Participants received migalastat 150 milligrams (mg) orally every other day (QOD) during the 12-week treatment period and the optional 36-week extension period.
Period: Treatment Period
Arm/Group | Migalastat
Started | 4
Safety Population (All enrolled participants who received at least 1 dose of study drug) | 4
Pharmacodynamics (PD) Population (Received study drug and had a non-missing baseline and postbaseline PD parameter recorded) | 4
Completed | 4
Not Completed | 0
Period: Extension Period
Arm/Group | Migalastat
Started | 4
Completed | 3
Not Completed | 1
Not completed — Low Compliance | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: all participants who received at least 1 dose of study drug.
Groups:
- Migalastat: Participants received migalastat 150 mg orally QOD during the 12-week treatment period and the optional 36-week extension period.
Arm/Group | Migalastat
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (21.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Who Experienced Severe Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as any adverse event with a start date on or after administration of study drug or pre-existing conditions that worsened on or after the start of the first study drug administration (on Day 1). A severe adverse event was defined as an adverse event that was incapacitating and required medical intervention. The number of participants who experienced one or more severe TEAEs after dosing on Day 1 through Week 48 is presented.
  A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Day 1 (after dosing) through Week 48 (end of extension period)
Population: Safety Population: all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Migalastat
Number analyzed (Participants) | 4
Participants | 1

2. Secondary Outcome: α-Galactosidase A (α-Gal A) Activity In Peripheral Blood Mononuclear Cells (PBMC) At Baseline, Week 12, And Week 48
Description: PBMCs were isolated from whole blood and lysed, and α-Gal A activity was measured by a validated fluorometric assay, with catalysis to fluorescent 4-methylumbelliferone (4-MU) as the activity measure. The activity values obtained were normalized to protein (measured using a colorimetric assay) and reported as enzyme activity (nanomole [nmol] 4-MU/hour [hr]) per mg of protein. On Day 1 of the first visit and at every visit thereafter, the samples were collected prior to dosing with migalastat.
  α-Gal A activity in PBMCs are presented by individual participants. Values of "0" presented below represent α-Gal A activity levels that were below the lower limit of quantification.
Time Frame: Baseline, Week 12 (end of treatment period), Week 48 (end of extension period)
Population: PD Population: All participants who received at least 1 dose of study drug and had at least 1 non-missing postbaseline PD parameter recorded. Participants who discontinued prior to the specified time point were not analyzed because no data were available.
Measure: Number; unit: nmol 4-MU/hr/mg protein
Arm/Group | Migalastat
Number analyzed (Participants) | 4
nmol 4-MU/hr/mg protein
  Participant 1 Baseline: number analyzed (Participants) | 1
  Participant 1 Baseline | 0.14
  Participant 1 Week 12: number analyzed (Participants) | 1
  Participant 1 Week 12 | NA — Data for this participant were below the limit of quantification.
  Participant 1 Week 48: number analyzed (Participants) | 1
  Participant 1 Week 48 | 0.12
  Participant 2 Baseline: number analyzed (Participants) | 1
  Participant 2 Baseline | 0.24
  Participant 2 Week 12: number analyzed (Participants) | 1
  Participant 2 Week 12 | 2.3
  Participant 2 Week 48: number analyzed (Participants) | 0
  Participant 3 Baseline: number analyzed (Participants) | 1
  Participant 3 Baseline | 0.21
  Participant 3 Week 12: number analyzed (Participants) | 1
  Participant 3 Week 12 | 2.43
  Participant 3 Week 48: number analyzed (Participants) | 0
  Participant 4 Baseline: number analyzed (Participants) | 1
  Participant 4 Baseline | 0.3
  Participant 4 Week 12: number analyzed (Participants) | 1
  Participant 4 Week 12 | 7.36
  Participant 4 Week 48: number analyzed (Participants) | 1
  Participant 4 Week 48 | 6.06

ADVERSE EVENTS:
Time Frame: Day 1 after dosing through Week 48 (end of extension period).
Arm/Group | Migalastat
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Migalastat (N=4)
Atrioventricular block (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Migalastat (N=4)
Atrial Fibrillation (Cardiac disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oedema Peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Bifascicular block (Cardiac disorders) | 1
Bundle branch block left (Cardiac disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Pain (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 1
QRS axis abnormal (Investigations) | 1
Venous pressure jugular increased (Investigations) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Nervousness (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1
Poor peripheral circulation (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can only publish the results from this trial provided they supply the sponsor (or authorized entity) a copy of any proposed publication for review. If requested, the investigator will remove information deemed confidential or proprietary by the sponsor and will withhold publication for an additional period of time to allow the sponsor to take appropriate measures to establish and preserve its proprietary rights.